CLINICAL TRIAL: NCT01974388
Title: Impact of Extent of Antral Resection on Surgical Outcomes of Sleeve Gastrectomy for Morbid Obesity (A Prospective Randomized Study)
Brief Title: Impact of Extent of Antral Resection on Outcomes of Sleeve Gastrectomy
Acronym: LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Ass. Prof., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Morbid Obesity
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
Keywords: Bariatric surgery, sleeve gastrectomy, gastric leak
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LSG started 2 cm from the pylorus (Active Comparator): laparoscopic sleeve gastrectomy starting 2 cm from the pylorus
  Interventions: Procedure: LSG started 2 cm from the pylorus
- LSG started 6 cm from pylorus (Active Comparator): LSG started 6 cm from pylorus
  Interventions: Procedure: LSG started 6 cm from pylorus

INTERVENTIONS:
Procedure: LSG started 2 cm from the pylorus — Laparoscopic sleeve gastrectomy started 2 cm from pylorus
  Other Names: Group I
  Arms: LSG started 2 cm from the pylorus
Procedure: LSG started 6 cm from pylorus — LSG started 6 cm from pylorus
  Other Names: Group II
  Arms: LSG started 6 cm from pylorus

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is a surgical technique that treats morbid obesity by both restrictive and hormonal action.

Consecutive patients with morbid obesity treated by LSG at our department were evaluated. Patients enrolled in the study were randomized into Group I: LSG begin the division 2 cm from the pylorus and Group II: LSG begin the division 6 cm from the pylorus. The primary outcome measure was the % of excess weight loss (%EWL); secondary outcomes included operative time, day to resume oral feeding, postoperative morbidity and mortality, improvement of comorbidity.

DETAILED DESCRIPTION:
This prospective randomized study was designed to compare between the beginning of sleeve gastrectomy 2 cm versus 6 cm from the pylorus with special regards to intraoperative problems, weight loss, improvement of comorbidities, postoperative complications, nutritional and elemental deficiencies.

Consecutive patients, who were treated for morbid obesity by laparoscopic sleeve gastrectomy (LSG) at the department of general surgery, Mansoura University, Egypt, during the period from January 2008 to January 2012, were eligible for the study. The exclusion criteria included patients above 60 or below 18 years old, history of upper laparotomy, unfit for anaesthesia or laparoscopy, major psychological instability, and drug abuse.

The operation was done under general anesthesia. Patient was in supine position with splitting of the operating table legs.Gastric transection started 2 cm proximal to the pylorus using 60 mm, green endo-stapler (Ethicon, USA) (GI) or 6 cm from the pylorus (G II). The following staplers were placed approximately 1 cm from the bougie in the direction of the gastroesophageal junction.

Group I: LSG begin the division 2 cm from the pylorus and Group II: LSG begin the division 6 cm from the pylorus. The primary outcome measure was the % of excess weight loss (%EWL); secondary outcomes included operative time, day to resume oral feeding, postoperative morbidity and mortality, improvement of comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* patients, who were treated for morbid obesity by laparoscopic sleeve gastrectomy (LSG)

Exclusion Criteria:

* patients above 60 or below 18 years old, history of upper laparotomy, unfit for anaesthesia or laparoscopy, major psychological instability, and drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
percent of excess weight loss | one year postoperative
  The percent of EWL was calculated as follows: [(preoperative weight-follow up weight)/preoperative excess weight] ×100.

SECONDARY OUTCOMES:
length of postoperative stay | 30 days
  length of postoperative stay
postoperative complications | one year postoperative
  gastric leakage, internal haemorrhage, pulmonary complications). Complications were graded according to their severity on a validated five point scale using Dindo-Clavien complication classification system) into (grades I, II, IIIa-b, IVa-b, V). Grade I (no need for specific intervention), grade II (need for drug therapy such antibiotics, blood transfusion, total parenteral nutrition), grade IIIa-b (need for invasive therapy radiological, endoscopic or surgical), grade IVa-b (organ dysfunction requiring ICU stay and management), grade V (death)
weight regain | one year postoperative
  an increase of body weight of more than 10 kg from the nadir
Resolution of comorbidity | one year postoperative
  Resolution of comorbidity was considered if the disease is controlled without any medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Study Director — Mansoura University
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Result] Ferrer-Marquez M, Belda-Lozano R, Ferrer-Ayza M. Technical controversies in laparoscopic sleeve gastrectomy. Obes Surg. 2012 Jan;22(1):182-7. doi: 10.1007/s11695-011-0492-0. PMID 21861236
- [Result] Pomerri F, Foletto M, Allegro G, Bernante P, Prevedello L, Muzzio PC. Laparoscopic sleeve gastrectomy--radiological assessment of fundus size and sleeve voiding. Obes Surg. 2011 Jul;21(7):858-63. doi: 10.1007/s11695-010-0255-3. PMID 20730606
- [Result] Shi X, Karmali S, Sharma AM, Birch DW. A review of laparoscopic sleeve gastrectomy for morbid obesity. Obes Surg. 2010 Aug;20(8):1171-7. doi: 10.1007/s11695-010-0145-8. PMID 20379795
- [Result] Sanchez-Santos R, Masdevall C, Baltasar A, Martinez-Blazquez C, Garcia Ruiz de Gordejuela A, Ponsi E, Sanchez-Pernaute A, Vesperinas G, Del Castillo D, Bombuy E, Duran-Escribano C, Ortega L, Ruiz de Adana JC, Baltar J, Maruri I, Garcia-Blazquez E, Torres A. Short- and mid-term outcomes of sleeve gastrectomy for morbid obesity: the experience of the Spanish National Registry. Obes Surg. 2009 Sep;19(9):1203-10. doi: 10.1007/s11695-009-9892-9. Epub 2009 Jul 2. PMID 19572113
- [Derived] Abdallah E, El Nakeeb A, Youssef T, Abdallah H, Ellatif MA, Lotfy A, Youssef M, Elganash A, Moatamed A, Morshed M, Farid M. Impact of extent of antral resection on surgical outcomes of sleeve gastrectomy for morbid obesity (a prospective randomized study). Obes Surg. 2014 Oct;24(10):1587-94. doi: 10.1007/s11695-014-1242-x. PMID 24728866
- See also: Mansoura university, Mansoura, Egypt — http://www.mans.edu.eg/